CLINICAL TRIAL: NCT04813848
Title: Effectiveness of a Bonding and a Fluoride Varnish for Long-term Dentin Hypersensitivity Treatment: a Split-mouth Randomized Clinical Trial
Brief Title: Effectiveness of a Bonding and a Fluoride Varnish for Long-term Dentin Hypersensitivity Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Livia Ottolenghi, DDS, PhD, Full Professor, Deputy Dean of the Faculty of Medicine and Dentistry, Dean of the Dental School, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5877/2020
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: To Decrease Dentin Hypersensitivity
Keywords: dentin hypersensitivity; bonding agent; fluoride varnish
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: A randomized, slit-mouth, double blind clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Varnish fluoride (Experimental): Varnish fluoride to be applied on the surface of exposed dentin
  Interventions: Procedure: Application of varnish fluoride desensitizing agent on buccal surfaces of exposed dentin
- Bonding agent (Active Comparator): Bonding agent to be applied on the surface of exposed dentin
  Interventions: Procedure: Application of bonding agent desensitizing agent on buccal surfaces of exposed dentin

INTERVENTIONS:
Procedure: Application of varnish fluoride desensitizing agent on buccal surfaces of exposed dentin — Varnish fluoride is a single dose transparent varnish with 5 % sodium fluoride (22.600 ppm fluoride) and 5 % calcium fluoride.
  The application was performed according to the manufacturer's instructions. The varnish was applied on a clean and dry surface, then after 10-20 seconds to allow the fluoride varnish to be absorbed, was then dried with air.
  Other Names: Bifluorid, Voco GmbH
  Arms: Varnish fluoride
Procedure: Application of bonding agent desensitizing agent on buccal surfaces of exposed dentin — Bonding agent is a single dose dual curing universal adhesive and its application was performed according to the manufacturer's instruction for cases with hypersensitive tooth necks. The bonding was applied without etching, on a clean and dry surface. After 10 s any excess material was removed and then light cured for 30 s.
  Other Names: Futurabond U, Voco GmbH
  Arms: Bonding agent

SUMMARY:
Objectives:

The aim of this in vivo randomized clinical trial with split-mouth design was to evaluate the clinical efficacy of one in-office application of a fluoride containing varnish and in office application of a bonding resin in adult patients presenting with dentin hypersensitivity.

Materials and Methods:

The study cohort consisted of 38 Caucasian outpatients, giving a total of 180 teeth were treated by fluoride varnish (FV) and 160 - by bonding agent (BA). Baseline pain in FV group was slightly higher on both scales (SCHIFF and VAS). Outcome measurements were assessed one or two weeks before product application (enrollment), at baseline at the application days (end of the run-in period: T0a, T0b, T0c), and at 1 week and at 1-2-6 months after first treatment.

ELIGIBILITY:
Inclusion Criteria:

* absence of systemic pathologies (ASA class I);
* not pregnant or lactating;
* good oral hygiene;
* with ≥1 sensitive tooth with exposed dentin on upper or lower dental arches;
* contemporary presence of exposed dentin both on the left and right counterpart of upper or lower arch.

Exclusion Criteria:

* domestic or in-office professional fluoride application and bleaching 6 months before beginning of treatment;
* long-term use of anti-inflammatory, analgesic and psychotropic drugs;
* eating disorders, systemic conditions that cause or predispose patients to develop dentin hypersensitivity (for example, Gastroesophageal reflux disease);
* periodontal surgery and within the previous three months before the study;
* orthodontic treatment within the previous three months before the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Level of Pain assessment with the Schiff Sensitivity Scale | All study participants were asked to record the pain intensity score at the baseline, before the application of the desensitizing agents
  A score of 0, 1, 2 or 3 was given by the participant. 0 = No subject response to stimulus, 1 = Subject response but will continue, 2 = Subject responds and moves or requests discontinuation, 3 = Painful response to stimulus, discontinuation requested.
  The lower the score, the lower the hypersensitivity. Air-blast stimulus was used: the response to a jet of cold air was rated by the examiner.
Level of Pain assessment with the Schiff Sensitivity Scale | All study participants were asked to record the pain intensity score at seven days after the application of the desensitizing agents
  A score of 0, 1, 2 or 3 was given by the participant. 0 = No subject response to stimulus, 1 = Subject response but will continue, 2 = Subject responds and moves or requests discontinuation, 3 = Painful response to stimulus, discontinuation requested.
  The lower the score, the lower the hypersensitivity. Air-blast stimulus was used: the response to a jet of cold air was rated by the examiner.
Level of Pain assessment with the Schiff Sensitivity Scale | All study participants were asked to record the pain intensity score at one month after the application of the desensitizing agents
  A score of 0, 1, 2 or 3 was given by the participant. 0 = No subject response to stimulus, 1 = Subject response but will continue, 2 = Subject responds and moves or requests discontinuation, 3 = Painful response to stimulus, discontinuation requested.
  The lower the score, the lower the hypersensitivity. Air-blast stimulus was used: the response to a jet of cold air was rated by the examiner.
Level of Pain assessment with the Schiff Sensitivity Scale | All study participants were asked to record the pain intensity score at two months after the application of the desensitizing agents
  A score of 0, 1, 2 or 3 was given by the participant. 0 = No subject response to stimulus, 1 = Subject response but will continue, 2 = Subject responds and moves or requests discontinuation, 3 = Painful response to stimulus, discontinuation requested.
  The lower the score, the lower the hypersensitivity. Air-blast stimulus was used: the response to a jet of cold air was rated by the examiner.
Level of Pain assessment with the Schiff Sensitivity Scale | All study participants were asked to record the pain intensity score at six months after the application of the desensitizing agents
  A score of 0, 1, 2 or 3 was given by the participant. 0 = No subject response to stimulus, 1 = Subject response but will continue, 2 = Subject responds and moves or requests discontinuation, 3 = Painful response to stimulus, discontinuation requested.
  The lower the score, the lower the hypersensitivity. Air-blast stimulus was used: the response to a jet of cold air was rated by the examiner.

SECONDARY OUTCOMES:
Level of Pain assessment with the Visual Analogue Scale (VAS) | All study participants were asked to record the pain intensity score at the baseline, before the application of the desensitizing agents
  The level of pain was evaluated on a visual scale from 0 ("no pain") to 10 ("maximum pain").
  The lower the score, the lower the hypersensitivity. Air-blast stimulus was used: the response to a jet of cold air was rated by the examiner.
Level of Pain assessment with the Visual Analogue Scale (VAS) | All study participants were asked to record the pain intensity score at seven days after the application of the desensitizing agents
  The level of pain was evaluated on a visual scale from 0 ("no pain") to 10 ("maximum pain").
  The lower the score, the lower the hypersensitivity. Air-blast stimulus was used: the response to a jet of cold air was rated by the examiner.
Level of Pain assessment with the Visual Analogue Scale (VAS) | All study participants were asked to record the pain intensity score at one month after the application of the desensitizing agents
  The level of pain was evaluated on a visual scale from 0 ("no pain") to 10 ("maximum pain").
  The lower the score, the lower the hypersensitivity. Air-blast stimulus was used: the response to a jet of cold air was rated by the examiner.
Level of Pain assessment with the Visual Analogue Scale (VAS) | All study participants were asked to record the pain intensity score at two months after the application of the desensitizing agents
  The level of pain was evaluated on a visual scale from 0 ("no pain") to 10 ("maximum pain").
  The lower the score, the lower the hypersensitivity. Air-blast stimulus was used: the response to a jet of cold air was rated by the examiner.
Level of Pain assessment with the Visual Analogue Scale (VAS) | All study participants were asked to record the pain intensity score at six months after the application of the desensitizing agents
  The level of pain was evaluated on a visual scale from 0 ("no pain") to 10 ("maximum pain").
  The lower the score, the lower the hypersensitivity. Air-blast stimulus was used: the response to a jet of cold air was rated by the examiner.

CONTACTS AND LOCATIONS:
Overall Officials: Livia Ottolenghi, DDS,PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Department of Oral and Maxillo-Facial Sciences, Sapienza University of Rome, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazur M, Jedlinski M, Ndokaj A, Ardan R, Janiszewska-Olszowska J, Nardi GM, Ottolenghi L, Guerra F. Long-Term Effectiveness of Treating Dentin Hypersensitivity with Bifluorid 10 and Futurabond U: A Split-Mouth Randomized Double-Blind Clinical Trial. J Clin Med. 2021 May 12;10(10):2085. doi: 10.3390/jcm10102085. PMID 34066300